CLINICAL TRIAL: NCT04698694
Title: Tolerability of Intramuscular Electroporation Delivery by Cliniporator® in Healthy Volunteers
Brief Title: ElectroPoration In a Clinical Setting
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Rottapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPIC trial
Record Dates: First submitted 2020-12-14; First posted 2021-01-07 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Tolerance
Keywords: coronavirus infection; vaccine; intramuscular electroporation
MeSH Terms: conditions — Coronavirus Infections | interventions — Electroporation

STUDY DESIGN:
Intervention Model Description: Twenty (20) subjects will be randomized 1:1 to one of the following EP conditions:
  1. voltage amplitude of 40 V (10 subjects)
  2. voltage amplitude of 60 V (10 subjects).
Who Masked: Participant, Investigator
Masking Description: The subjects and investigators will remain blind with respect to the voltage strength received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects treated with Cliniporator® using a voltage amplitude of 40 V (Experimental): 10 subjects deemed eligible are between 18-55 y of age respected the inclusion and exclusion criteria will be selected in a randomized way (1:1) and treated with a voltage amplitude of 40 V.
  Interventions: Device: Electroporation with voltage amplitude of 40 V (corresponding to an electric field strength of 100 V/cm)
- Subjects treated with Cliniporator® using a voltage amplitude of 60 V (Experimental): 10 subjects deemed eligible are between 18-55 y of age respected the inclusion and exclusion criteria will be selected in a randomized way (1:1) and treated with a voltage amplitude of 60 V.
  Interventions: Device: Electroporation with voltage amplitude of 60 V (corresponding to an electric field strength of 150 V/cm)

INTERVENTIONS:
Device: Electroporation with voltage amplitude of 40 V (corresponding to an electric field strength of 100 V/cm) — The physician will select the voltage amplitude of 40 V to be given to the subject based on a randomization list, while the subject will remain blind to the voltage he/she is assigned to. The electroporation will be performed with a EPS electrode gun.
  Arms: Subjects treated with Cliniporator® using a voltage amplitude of 40 V
Device: Electroporation with voltage amplitude of 60 V (corresponding to an electric field strength of 150 V/cm) — The physician will select the voltage amplitude of 60 V to be given to the subject based on a randomization list, while the subject will remain blind to the voltage he/she is assigned to. The electroporation will be performed with a EPS electrode gun.
  Arms: Subjects treated with Cliniporator® using a voltage amplitude of 60 V

SUMMARY:
This is a single-blind, single-center, randomized, study in healthy subjects in which the volunteer patients will remain blind with respect to the voltage strength received.

DETAILED DESCRIPTION:
Background:

The major obstacle to the preventive or therapeutic success of DNA vaccines is undoubtedly their delivery. If this cannot be made simple, cheap and effective, they may not become a viable option for human use. Numerous clinical trials have confirmed that a standard needle and syringe parenteral (mainly intramuscular or intradermal) delivery is not enough. An important tenet, confirmed by different DNA immunization studies, is that electroporation dramatically enhances the expression of the encoded antigen as well as the potency and immunogenicity of DNA vaccines. Electroporation (EP) creates transient increases in cell membrane permeability, thus enhancing DNA uptake and leading to a more robust immune response. EP involves the application of brief electric pulses to tissue in order to permeabilize cell membranes in a transient and reversible manner. The temporary formation of pores facilitate successful transport of macromolecules, like DNA, that occurs on the order of microseconds vs. minutes in the case of passive diffusion alone. EP is considered a safe and well validated procedure that can easily be handled as an out-patient procedure. In this regard, electrochemotherapy and electro gene transfer with the Cliniporator® (IGEA Srl, Carpi, Italy) has been added to clinical practice.

Aim of the present study is therefore to formally confirm the tolerability of electroporation given by the EPSGT gun and the Cliniporator® device in a clinical setting of healthy volunteers, prior to the phase I/II study of the COVID-19 vaccine in a similar population.

Study Design:

Twenty (20) subjects will be randomized 1:1 to one of the following EP conditions:

1. voltage amplitude of 40 V (10 subjects)
2. voltage amplitude of 60 V (10 subjects). For the purpose of the study, 0.5 ml of sterile 0.9% saline solution will be injected intramuscularly into the deltoid muscle of the right arm using a common insulin syringe inserted in the EPS gun; the saline injection will immediately be followed by electroporation given by the gun connected to the electrical pulse generator, Cliniporator®.

The electroporation technology has been optimized by IGEA developing a dedicated EPS electrode gun. The EPS gun is an intuitive and handful procedure that combines in the same device the injection of a DNA vaccine (or a sterile 0.9% saline solution as in the case of the present study) and the delivery of the electrical pulses; the procedure is completed in few seconds. The EP needles 7 (diameter 0.45 mm) are hidden under a sliding cap integrated into the EPS gun, to reduce perceived pain potentially associated to anxiety or fear. The EPS gun allows the insertion of both the electrode needles and the syringe needle into the muscle. By pressing the syringe plunger, the content of the syringe will be injected, by pulling the trigger the syringe needle will be retracted, and finally the electrical pulses will be delivered by pressing a pedal connected to the pulse generator.

Pain assessment:

On the day of injection and EP, subjects will be instructed to measure the length of time pain is experienced by using a stopwatch. Additionally, subjects will complete the Visual Analog Scale (VAS) to rate the level of pain experienced immediately (0 min) and after 5 min, 15 min, 30 min, and 60 min post-EP. In addition subjects will rate discomfort level using an 11-point numerical rating scale (NRS), evaluated 60' (T4) after the procedure. On Day 2 and Day 7 post-EP, subjects will complete again the VAS as described above, and NRS. In addition, on Day 1 (T2, +15'), Day 2 and Day 7 subjects will complete a self-administered questionnaire assessing the acceptance of the procedure. Therefore, to better measure the acceptability of the injection related to the use of a new device from people's own perspectives, all participants will complete the Perception of Injection (PIN) questionnaire, adapted from the Vaccines' Perception of Injection (VAPI) questionnaire.

Safety Analysis:

Safety analyses will include summaries of the following:

* adverse events, including severity and relationship to the procedure (to the intramuscular injection, to the electroporation, or to both procedures)
* serious adverse events, including severity and relationship to the procedure (to the intramuscular injection or to the electroporation, or to both)
* abnormal changes in CPK
* abnormal changes in vital signs and ECG

Sample size and Statistical Analysis:

No sample size calculation was performed on this study on the tolerability of two EP voltage strengths.

The statistical analyses will be mainly descriptive. Qualitative variables will be summarized by counts and percentages, while quantitative characteristics by quartiles or mean and standard deviation, as appropriate.

Data collected longitudinally will be also described appropriately. Specific summary indices will be calculated on the longitudinal VAS profiles (e.g. SPID and peak PID) and the agreement between VAS and NRS collected at each time point will be also assessed.

All adverse events will be graded in accordance with the 2007 FDA toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening) and will be reported as percentages and narratives will be also presented.

Study Management:

The data requested by the study will be reported in an electronic remote data capture system (e-CRF). The subject data collected in the e-CRF during the study will be documented anonymously and the subject can only be identified by an identification code.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before undergoing any study-specific procedure
2. Healthy subjects, as determined by a responsible physician, based on a medical evaluation including medical history and physical examination
3. Males or females aged ≥18 and ≤ 55 years
4. A minimum weight of 50 kg and Body Mass Index >18.5 and ≤30 kg/m2
5. Vital signs within the following values or ranges:

   1. Body temperature ≤ 37,5 °C
   2. Pulse frequency ≥51 and ≤100 beats per minute
   3. Diastolic BP ≥60 mmHg, ≤ 90 mmHg
   4. Systolic BP ≥ 90 mmHg, ≤ 140 mmHg
6. Normal ECG
7. CPK within normal reference range
8. Non-pregnant women of childbearing potential, non-breastfeeding
9. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. Any past or present cardiac disease, even if not evident at ECG
2. Bleeding disorders (e.g. coagulopathy or platelet disorder or coagulation factor deficiency) or prior history of significant bleeding or bruising following IM injections or venepuncture
3. History of seizures or mental illness
4. Metal implants within 20 cm of the planned site(s) of injection
5. Presence of keloid scar formation or hypertrophic scar, or other clinically significant medical condition at the planned site(s) of injection
6. Any abnormality or permanent body art (e.g. tattoos) that would interfere with the ability to observe local reactions at the injection site in the deltoid area
7. History of alcohol or drug abuse during the 12 months preceding the screening
8. Pregnancy (i.e. positive pregnancy test) or willingness/intention to become pregnant during the study
9. Breastfeeding
10. Any other clinically relevant disease and condition that, in the opinion of the Investigator, may jeopardize efficacy or safety assessments or may compromise the subject's safety during trial participation.

Ages: 18 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Pain of intramuscular delivery of a sterile solution followed by electroporation | approximately 1 month
  Subjsects will rate the intramuscolar pain using the Visual Analog Scale (VAS) to rate the level of pain experienced from the minimum value of "No Pain" and the maximum value "Pain as bad as it could possibly be".
Discomfort level of intramuscular delivery of a sterile solution followed by electroporation | approximately 1 month
  Subjsects will rate discomfort level using an 11-point Numerical Rating Scale (NRS). Scores range from the minimum value 0 that means ''None'' to 10 that means ''Severe''.
Pain of intramuscular delivery of a sterile solution followed by electroporation | approximately 1 month
  Subjsects will rate the Perseption of Injection (PIN) questionnaire. Scores range from the minimum value 1 that means ''None'' to 5 that means ''very very much''.

SECONDARY OUTCOMES:
Incidence of Injection site Adverse Events | approximately 1 month
  Number of AE at the injection site
Incidence of sistemic Adverse Events | approximately 1 month
  Number of sistemic AE

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza-Ospedale San Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frelin L, Brass A, Ahlen G, Brenndorfer ED, Chen M, Sallberg M. Electroporation: a promising method for the nonviral delivery of DNA vaccines in humans? Drug News Perspect. 2010 Dec;23(10):647-53. doi: 10.1358/dnp.2010.23.10.1513492. PMID 21180650
- [Background] Mir LM. Application of electroporation gene therapy: past, current, and future. Methods Mol Biol. 2008;423:3-17. doi: 10.1007/978-1-59745-194-9_1. PMID 18370187
- [Background] Paul-Dauphin A, Guillemin F, Virion JM, Briancon S. Bias and precision in visual analogue scales: a randomized controlled trial. Am J Epidemiol. 1999 Nov 15;150(10):1117-27. doi: 10.1093/oxfordjournals.aje.a009937. PMID 10568628
- [Background] Rizzuto G, Cappelletti M, Maione D, Savino R, Lazzaro D, Costa P, Mathiesen I, Cortese R, Ciliberto G, Laufer R, La Monica N, Fattori E. Efficient and regulated erythropoietin production by naked DNA injection and muscle electroporation. Proc Natl Acad Sci U S A. 1999 May 25;96(11):6417-22. doi: 10.1073/pnas.96.11.6417. PMID 10339602